CLINICAL TRIAL: NCT02171026
Title: Relative Bioavailability of Dabigatran and Amiodarone After Multiple Oral Administrations of 150 mg Dabigatran Etexilate b.i.d. With or Without 600 mg Amiodarone as Single Dose in Healthy Male and Female Volunteers (an Open-Label, Multiple-Dose, Group-Comparison Study)
Brief Title: Bioavailability of Dabigatran and Amiodarone After Multiple Oral Administrations of Dabigatran Etexilate With or Without Amiodarone as Single Dose in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.57
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Amiodarone

ARMS (2):
- Dabigatran etexilate + Amiodarone (Experimental)
  Interventions: Drug: Dabigatran etexilate; Drug: Amiodarone
- Amiodarone (Active Comparator)
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Dabigatran etexilate
  Arms: Dabigatran etexilate + Amiodarone
Drug: Amiodarone

SUMMARY:
Investigation of the bioavailability, safety and tolerability of dabigatran with and without concomitant administration of amiodarone and the bioavailability of amiodarone and desethylamiodarone after administration of a single dose of amiodarone with and without dabigatran

ELIGIBILITY:
Inclusion Criteria:

Healthy males and females according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (BP, pulse rate (PR)), 12-lead ECG, clinical laboratory tests
2. Aged >=18 and <=55 years
3. Body mass index (BMI) >=18.5 and BMI <=29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study according to GCP and local legislation

Exclusion Criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. Diseases of the central nervous system, such as epilepsy; psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity, including drug allergy, which was deemed relevant to the study as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the study
9. Use of drugs, which might have reasonably influenced the results of the study based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the study
10. Participation in another study with an investigational drug within two months prior to administration or during the study
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation; more than 100 mL within four weeks prior to administration or during the study
14. Excessive physical activities; within one week prior to administration or during the study
15. Any laboratory value outside the reference range that was of clinical relevance
16. Inability to comply with dietary regimen of study centre
17. Females of child bearing potential who were pregnant, breast feeding or who were either not surgically sterile or were sexually active and not using an acceptable, i.e. highly effective with a Pearl index >1%, form of contraception as either the oral contraceptives since at least two months and the double barrier method, i.e. intrauterine device with spermicide and condom for the male partner 18.) Male subjects had to agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post-study medical. Acceptable methods of contraception comprised barrier contraception and a medically accepted contraceptive method for the female partner (intrauterine device with spermicide, hormonal contraceptive since at least two month).

19.) Abnormal thyroid stimulating hormone (TSH) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-04; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration time curve of the analyte in plasma over one steady state dosing interval) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h post-dose on day 3, pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose on day 4
Cmax,ss (maximum concentration of the analyte in plasma at steady state) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h post-dose on day 3, pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose on day 4
AUC0-infinity (area under the concentration time curve of the analyte in plasma extrapolated to infinity) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
Cmax (maximum concentration of the analyte in plasma) | pre-dose on day 1 and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
Changes in aPTT (activated partial thromboplastin time) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
Changes in ECT (ecarin clotting time) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
AUERτ,ss (area under the effect ratio-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
ERmax,ss (maximum effect ratio in plasma at steady state) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose

SECONDARY OUTCOMES:
AUC0-tz,ss (area under the concentration-time curve of the analyte in plasma from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
tz,ss (time of last measurable concentration of the analyte in plasma within the dosing interval τ at steady state) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
tmax,ss (time from last dosing to the maximum concentration of the analyte in plasma at steady state on Day 4) | pre-dose Day 4 and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
CL/Fss (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
CLR,ss (renal clearance of the analyte at steady state determined over the dosing interval τ) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
tmin,ss (time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
Cpre,ss (pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
MRTp.o.,ss (mean residence time of the analyte in the body at steady state after oral administration) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
Vz/Fss (apparent volume of distribution of the analyte during the terminal phase λz at steady state following an extravascular administration) | pre-dose on Day 1, 2, 3, and 4; on day 3 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h post-dose; on day 4 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 h post-dose
Aeτ,ss (amount of the analyte eliminated in urine at steady state over an uniform dosing interval τ) | pre-dose, 0-12 h and 12-24 h post-dose on days 3 and 4
feτ,ss (fraction of the analyte eliminated in urine at steady state over a uniform dosing interval τ) | pre-dose, 0-12 h and 12-24 h post-dose on days 3 and 4
AUC 0-tz (area under the concentration-time curve of the analyte in plasma over the time interval 0 to the last quantifiable analyte plasma concentration after single dose administration) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
tz (time of last measurable concentration of the analyte in plasma following a single dose) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
%AUCtz-infinity (percentage of the AUC0-infinity of the analyte obtained by extrapolation) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
tmax (time from dosing to the maximum concentration of the analyte in plasma following a single dose) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
λz (terminal rate constant of the analyte in plasma after a single dose) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
t1/2 (terminal half-life of the analyte in plasma after a single dose) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
MRTp.o. (mean residence time of the analyte in the body after single dose p.o. administration | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
CL/F (apparent clearance of the analyte in the plasma after extravascular single dose administration) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
Vz/F (apparent volume of distribution of the analyte during the terminal phase λz following extravascular dose) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96 and 120 h post-dose
Changes in physical examination | up to 8 days following drug administration
Changes in vital signs (BP, PR) | up to 8 days following drug administration
Changes in 12-lead electrocardiogram (ECG) | up to 8 days following drug administration
Changes in clinical laboratory tests | up to 8 days following drug administration
Occurrence of adverse events | up to 8 days following drug administration
Assessment of tolerability by investigator | up to 8 days following drug administration